CLINICAL TRIAL: NCT01571908
Title: Rapid Sequence Intubation With Magnesium-rocuronium Compared With Succinylcholine - A Randomised Clinical Study
Acronym: MagInRoc
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Christoph Czarnetzki, Responsable Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CER 11-235
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-05

CONDITIONS: Intubation Conditions
Keywords: rocuronium; succinylcholine; magnesiumsulphate; intubation conditions
MeSH Terms: interventions — Magnesium; Rocuronium; Sodium Chloride; Succinylcholine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium perfusion - Rocuronium (Experimental): 60 mg/kg of magnesium perfusion over 15 minutes before Anaesthesia. After Anaesthesia induction 0.6 mg/kg of Rocuronium intravenously
  Interventions: Drug: Magnesium perfusion; Drug: Rocuronium
- Placebo perfusion - Succinylcholine (Active Comparator): 1ml/kg of saline (placebo) over 15 minutes before Anaesthesia. After Anaesthesia induction 1 mg/kg of Succinylcholine intravenously
  Interventions: Drug: Placebo perfusion; Drug: Succinylcholine

INTERVENTIONS:
Drug: Magnesium perfusion — The patient receives during 15 minutes a perfusion of 60mg/kg of Magnesium sulphate before induction of anaesthesia.
  Other Names: Magnesium
  Arms: Magnesium perfusion - Rocuronium
Drug: Rocuronium — Immediately after anaesthesia induction and loss of consciousness 0,6 mg/kg of rocuronium will be injected
  Other Names: Zemuron
  Arms: Magnesium perfusion - Rocuronium
Drug: Placebo perfusion — The patient receives during 15 minutes a perfusion of 1 ml/kg of saline before induction of anaesthesia
  Other Names: Saline
  Arms: Placebo perfusion - Succinylcholine
Drug: Succinylcholine — Immediately after anaesthesia induction at loss of consciousness 1 mg/kg of succinylcholine will be injected
  Other Names: Anectine
  Arms: Placebo perfusion - Succinylcholine

SUMMARY:
Magnesium accelerates the reaction of rocuronium, a neuromuscular blocker used for muscle relaxation to ease the intubation during anaesthesia.

Succinylcholine is a very fast reacting neuromuscular blocker. It is often used in emergency procedures, when rapid intubation is necessary.

We want to now if a perfusion of magnesium before anaesthesia accelerates to such an extent the reaction of rocuronium that intubation conditions are comparable or even better than with succinylcholine alone (prior perfusion of saline=placebo)

DETAILED DESCRIPTION:
Rapid sequence intubation (RSI) is the preferred method of endotracheal intubation in the emergency setting. The aim of RSI is to achieve rapid unconsciousness and complete neuromuscular blockade which facilitates endotracheal intubation. RSI is of particular importance in unfastened patients who are at risk of regurgitation and subsequent aspiration of stomach contents into the lungs during induction of anaesthesia.

Still today, succinylcholine is the neuromuscular blocking agent of choice for RSI. However, unfortunately in 60 at 80% the intubations conditions not are excellent and there are contraindications for the usage of succinylcholine and numerous side effects. Thus there is a need for alternative techniques that allow for rapid, high-quality and safe intubation conditions. Magnesium has an impact on neuromuscular transmission; it reduces the amount of acetylcholine that is released at the motor nerve terminal.

It has been shown that an IV infusion of magnesium sulphate prior to a standard intubation dose of rocuronium enhanced the speed of onset of the neuromuscular block compared with rocuronium alone by about 35% and there was much less variability in onset times. This makes the combination magnesium-rocuronium a potentially interesting alternative to succinylcholine for RSI.

The investigators objective is to compare in surgical patients during a standardized RSI procedure intubation conditions with rocuronium 0.6 mg kg-1 after pre-treatment with intravenous MgSO4 60 mg kg-1 (experimental intervention) with succinylcholine 1 mg kg-1 (control intervention) and to quantify any minor or major adverse event.

The investigators primary hypothesis is that with rocuronium 0.6 mg kg-1, after pre-treatment with MgSO4 60 mg kg-1, the rate of excellent intubation conditions will be higher (80%) compared with succinylcholine 1 mg kg-1 (60%).

This is a two centre (Division of Anaesthesiology, Geneva University Hospitals and Division of Anaesthesiology, University Hospital of Lausanne), stratified (male, female), randomized, double blinded study including 280 patients.

The investigators will compare in surgical patients during a standardized RSI procedure intubation conditions with rocuronium 0.6 mg kg-1 after pre-treatment with intravenous MgSO4 60 mg kg-1 (experimental intervention) with succinylcholine 1 mg kg-1 (control intervention).

Intubation conditions will be evaluated by the intubating anaesthesiologist following predefined criteria. The intubating anesthetist will not be present at study drug administration to guarantee blinding. Only two intubating anaesthetists will be identified per participating centre.

Rapid sequence intubation is a cornerstone of daily anaesthetic practice and succinylcholine is still the most frequently used neuromuscular agent in this context. In some patients, succinylcholine is contraindicated and therefore alternatives to this very fast reacting neuromuscular blocker are needed. If the investigators show that the investigators proposed magnesium-rocuronium regimen provides better intubation conditions as succinylcholine, the investigators study is likely to have an important impact on daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult, age ≥18 to 65 years, male or female.
* American Society of Anaesthesiology [ASA] status I or II.
* Patient is able to read and understand the information sheet and to sign and date the consent form.
* Patient scheduled of elective surgery lasting ≥60 minutes.
* If the patient is female and of childbearing potential, she must have a negative pregnancy test.

Exclusion Criteria:

* A history of allergy or hypersensitivity to rocuronium, succinylcholine or magnesium sulphate
* Neuromuscular disease
* History of malignant hyperthermia
* Preoperative medications known to influence neuromuscular function (for instance, certain antibiotics [aminoglycosides], anticonvulsants [phenytoine], or IV lidocaine)
* Electrolyte abnormalities* (for instance, hypermagnesemia or hyperkalemia)
* Hepatic dysfunction* (i.e. bilirubin >1.5 x upper limit normal (ULN), alanine aminotransferase (ALT) >2.5 x ULN, aspartate aminotransferase (AST) >2.5 x ULN)
* Renal insufficiency* (i.e. creatinine >1.5 x ULN, creatinine clearance < 60 ml min-1 1.73 m-2, estimated by the formula by Cockcroft-Gault)).
* Atrioventricular heart block
* Patients with magnesium treatment
* Patients with a body mass index <19 or >28 kg m2
* Pregnant or breastfeeding women
* Expected difficult intubation or mask ventilation.
* Patient having participated in any clinical trial within 30 days, inclusive, of signing the informed consent form of the current trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Intubation score | Patient will be followed over 24 hours
  Intubation conditions will be evaluated using a published score that takes into account ease of laryngoscopy (easy, fair, difficult), vocal cords position (abducted, intermediate/moving, closed) and presence of diaphragmatic movement or coughing while inserting the tube (none, slight, vigorous/sustained). The final score summarises intubation conditions as excellent (all qualities are excellent), good (all qualities are either excellent or good), or poor (presence of a single quality listed under "poor").

SECONDARY OUTCOMES:
Signs of histamine release | From start of anesthesia induction upto 30 minutes after intubation
  Immediately after intubation, patients will be evaluated for signs of histamine release (bronchospasm, erythema, oedema).
awareness and muscle pain | 24 hour follow up
  The day after surgery, patients will be visited and will be screened for awareness and muscle pain.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Czarnetzki, MD, PD, Principal Investigator — University hospitals of Geneva; Martin R Tramèr, MD, PhD, Study Chair — University hospitals of Geneva; Christian Kern, MD, Prof, Principal Investigator — University Hospitals of Lausanne, Switzerland
Locations (2):
- Switzerland (2):
  - University Hospital of Geneva, Anesthesia Department, Geneva, Canton of Geneva
  - Division of Anaesthesiology, University Hospital of Lausanne (CHUV), Lausanne, Canton of Vaud

REFERENCES:
- [Derived] Czarnetzki C, Albrecht E, Masouye P, Baeriswyl M, Poncet A, Robin M, Kern C, Tramer MR. Rapid Sequence Induction With a Standard Intubation Dose of Rocuronium After Magnesium Pretreatment Compared With Succinylcholine: A Randomized Clinical Trial. Anesth Analg. 2021 Dec 1;133(6):1540-1549. doi: 10.1213/ANE.0000000000005324. PMID 33337797